CLINICAL TRIAL: NCT01335828
Title: "ShearWave" Elastography Interest in the Management of Thyroid Nodules
Brief Title: Elastography Interest in the Management of Thyroid Nodules
Acronym: SWETHY
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AdministrateurCIC (Other)
Responsible Party: Sponsor-Investigator, AdministrateurCIC, principal investigator, University Hospital, Grenoble
Organization: University Hospital, Grenoble (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DCIC 10 24
Record Dates: First submitted 2010-11-10; First posted 2011-04-14 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Thyroid Nodules
Keywords: Echography; Elastography; Thyroid nodules; Needles punction; Thyroid surgery; Patients with thyroids nodules
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- echography/elastography (Other)
  Interventions: Device: Medical ultrasound device (ShearWave system)

INTERVENTIONS:
Device: Medical ultrasound device (ShearWave system) — Echography (all modes) and elastography "ShearWave" system

SUMMARY:
Define an ultrasound/elastography benignity criteria in strategy management of a patient population carries one or more thyroid nodules.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 years old
* Patient affiliated to social security or similarly regime
* Patients referred for fine needle aspiration or surgery with one or more thyroid nodules

Exclusion Criteria:

* Patients with too much thyroid nodules or topography too imprecise to allow unambiguous correlation between echo/elastography data and histology/cytology data
* Patients withan echography/elastography indications cons
* Pregnant women and lactating mothers
* Adult unable to express their consent
* Ward of court or under guardianship
* Person under legal protection
* Person deprived of freedom by judicial or administrative decision
* Person hospitalized without their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2010-11; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Defined echo/elastography benignity criteria | two and half years
  For ultrasound and elastography benignity criteria which will be retained, outcome focus on cytoponctions number for benin nodules can be avoided by taking into account this benign criteria

SECONDARY OUTCOMES:
Evaluate the diagnostic performance of elastography ShearWave for characterization of thyroid nodules in a population of patients referred for needle biopsy or surgery nodule thyroid | two and half years
  ROC curves for performance of ultrasound, elastography and their coupling, compared to the reference cytology / histology.
Assessing the use of elastography in clinical practice | two and half years

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Investigation Center - Technological Innovation - Inserm 803 - University Hospital France, Grenoble, France